CLINICAL TRIAL: NCT00963092
Title: Stomach and Oesophageal Cancer Study (SOCS)
Brief Title: Study of Blood and Tissue Samples From Patients With Stomach Cancer, Esophageal Cancer, or Gastroesophageal Junction Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CRUK-UC-SOCS-03-5-064; CDR0000636974 (Registry Identifier: PDQ (Physician Data Query)); EU-20911
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-07

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer; Gastric Cancer
Keywords: adenocarcinoma of the gastroesophageal junction; recurrent gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus; recurrent esophageal cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; stage IA gastric cancer; stage IB gastric cancer; stage IIA gastric cancer; stage IIB gastric cancer; stage IIIA gastric cancer; stage IIIB gastric cancer; stage IIIC gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Microarray Analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: microarray analysis
Genetic: protein analysis
Other: cytology specimen collection procedure
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Collecting and storing samples of tissue, blood, and saliva from patients with cancer to test in the laboratory may help the study of cancer in the future.

PURPOSE: This research study is collecting blood and tissue samples from patients with stomach cancer, esophageal cancer, or gastroesophageal junction cancer, studying them in the laboratory, and storing them for future studies.

DETAILED DESCRIPTION:
OBJECTIVES:

* To set up a population-based gastric and esophageal cancer cohort with comprehensive epidemiological, clinical, and pathological data in order to identify novel genetic and environmental risk factors for these cancers using an association study design.
* To establish a blood-based epidemiological resource with parallel tumor samples on a population-based series of gastric and esophageal cancer cases.
* Compare any differences in genetic susceptibility genes according to the site of esophago-gastric cancer (e.g., distal gastric, proximal gastric, or junctional and esophageal tumors) and the histopathological sub-type.
* Test existing molecular hypotheses and determine whether common genetic variants in candidate genes predispose to gastric and esophageal cancer by comparing the frequency of variants in cancer patients with that in controls.
* Generate new hypotheses of genetic and certain environmental determinants, explore the potential impact on cancer disease risk of a range of environmental factors that can be measured in plasma (e.g., antibodies to various infective agents, markers of systemic inflammation, markers of oxidation), and examine gene-environment interactions.
* Refine our understanding of risk factors that are identified (e.g.,chronic Helicobacter pylori infection and smoking) and examine how these interact with genetic determinants of disease.
* Define the proportion of gastric cancer incidence attributable to mutations in known predisposing genes, such as E-cadherin.
* Obtain data on molecular profiles of tumors (mostly paraffin-embedded, rarely frozen) using dense array technologies, therefore enabling studies of the interaction between germline polymorphisms and tumor somatic genotype upon tumor behavior, response to treatment, and patient outcome.

OUTLINE: This is a multicenter study.

Patients and healthy controls complete an epidemiological questionnaire, provide a blood sample for plasma and genetic analyses, and may also provide a saliva sample. Tumor samples (in the form of paraffin block material or, in rare cases, frozen) may also be obtained from the hospital where the patient underwent surgery.

White blood cells are assayed for DNA/RNA isolation to look at genetic variants. DNA is extracted from saliva to look at genetic variants. Plasma/serum samples are analyzed to look at proteins and serological markers. Tumor samples are used to review the histology type. Nucleic acids are extracted from tumor sample sections; retrieval of a small (0.6 mm) core from each section is used to construct a tissue microarray which are be analyzed by immunohistochemistry and FISH.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

PROJECTED ACCRUAL: A total of 1,000 patients per cancer (gastric and esophageal) and 2,000 controls will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must meet 1 of the following criteria:

  * Diagnosis of gastric or esophageal adenocarcinoma

    * Diagnosed within the past 5 years
    * May include gastro-esophageal junction tumor
  * Spouse or relative of the patient
  * Samples collected from the European Prospective Investigation of Cancer (EPIC) study
* Patients will be approached to participate in the study regardless of their current treatment being curative or palliative, medical or surgical, or if they are currently having follow-up clinical appointments

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2002-08; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Creation of repository of blood, saliva, and tumor samples

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Caldas, Principal Investigator — Cancer Research UK
Locations (1):
- Cancer Research UK at Cambridge Research Institute, Cambridge, England, United Kingdom